CLINICAL TRIAL: NCT04130555
Title: Observational Prospective Study of a Non-cross-linked Porcine Acellular Dermal Matrix in Ventral Mesh Rectopexy
Brief Title: Safety and Performance Evaluation of a Biological Matrix Used for Rectal Prolapse Repair by Ventral Rectopexy
Status: Completed | Type: Observational
Sponsor: Meccellis Biotech (Industry)
Responsible Party: Sponsor
Other Study IDs: RPR_01_CIP; 2019-A02024-53 (ID-RCB) (Other: ANSM)
Record Dates: First submitted 2019-10-14; First posted 2019-10-17 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Rectal Prolapse
Keywords: ventral rectopexy; biological mesh
MeSH Terms: conditions — Rectal Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CELLIS Rectopexy: Rectal prolapse repair by ventral rectopexy with the CELLIS Rectopexy matrix
  Interventions: Device: CELLIS Rectopexy (Porcine Acellular Dermal Matrix, PADM)

INTERVENTIONS:
Device: CELLIS Rectopexy (Porcine Acellular Dermal Matrix, PADM) — Biological membrane used in Laparoscopic Ventral Rectopexy (LVR) or robotic assisted rectopexy

SUMMARY:
The general objective of the study is to confirm the medium/long-term safety and clinical performance of the CELLIS Rectopexy membrane used in rectal prolapse repair by ventral rectopexy and to identify emerging risks in comparison to the clinical data related to other types of fixation material.

The present study will be a prospective multicentric non-randomized and non-controlled trial involving 55 patients followed for 24 months. The study will be conducted in France in 3 investigational centres.

DETAILED DESCRIPTION:
The study will be prospective, multicentric, single-arm, observational (non-interventional) to evaluate the safety and performance of CELLIS Rectopexy used in rectal prolapse repair by ventral rectopexy.

All evaluations will be performed and products used according to the usual practice, without additional or unusual diagnostic, treatment and monitoring procedure.

The study will be conducted in France in 3 investigational centres including 55 patients scheduled for the repair of rectal prolapse.

Each patient will participate in one assessment period including a screening visit, followed by the day of surgical procedure and a hospitalization period. Patients will return for ambulatory visits at Day 30 (+/- 7 days), Month 6 (+/- 2 weeks), Month 12 (+/- 2 weeks) and Month 24 (+/-2 weeks).

The surgical technique used to repair rectal prolapse will be either Laparoscopic Ventral Rectopexy (LVR) or a robotic assisted rectopexy with the use of the da Vinci Surgical System (Intuitive Surgical, Inc., Sunnyvale, CA).

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥18 years,
* Patient with an indication of rectal prolapse repair by ventral rectopexy (external and internal rectal prolapse),
* Patient being informed of its participation to the study and of the follow-up visits, and having no objection to the clinical data collection and medical file access,
* Patient being informed of the porcine origin of the device in advance of the procedure.

Exclusion Criteria:

* Patient with known hypersensitivity to porcine materials,
* Patient with an existing infection not appropriately treated,
* Patient who are pregnant,
* Patient having refused to participate to the study,
* Patient refusing to come back to the follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Constitution and follow-up of a consecutive cohort of patients operated with the CELLIS Rectopexy membrane based on the usual practices, the indication and the inclusion-exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Rate of adverse events including reoperation and removal of the mesh | From the surgical procedure through the entire 24-month follow-up period
  Percentage

SECONDARY OUTCOMES:
Rate of structural defect recurrence based on rectal examination with/without adjunctive investigations as clinically indicated | Throughout the study until end of the 24-month follow-up period
  Percentage
Rate of structural defect recurrence requiring reoperation | Throughout the study until end of the 24-month follow-up period
  Percentage
Symptoms evolution: presence or absence of symptoms (constipation, fecal incontinence, bloody and/or mucous rectal discharge (soiling), unsatisfactory sexual activity, pain) | At baseline and at 30-day, 6-month, 12-month and 24-month follow-up visits
  Described at each visit and compared to baseline
Symptoms severity scored by a visual analog scale (0-10; 0 corresponding to no impact on life and 10 corresponding to extreme, incapacitating impact) | At baseline and at 30-day, 6-month, 12-month and 24-month follow-up visits
  Described at each visit and compared to baseline
Rate of symptoms recurrence | Throughout the study until end of the 24-month follow-up period
  Percentage
Severity of disease by the use of the Cleveland Clinic Incontinence Score (CCIS) | At baseline and at 30-day, 6-month, 12-month and 24-month follow-up visits
  Change from screening of total score at each follow-up visit. This scoring system cross-tabulates frequencies and different anal incontinence presentations (Gas/Liquid/Solid/Pad use/Need for lifestyle alterations) and sums the returned score to a total of 0-20 (where 0 = perfect continence and 20 = complete incontinence).
Severity of disease by the use of the Obstructed Defecation Score (ODS) | At baseline and at 30-day, 6-month, 12-month and 24-month follow-up visits
  Change from screening of total score at each follow-up visit. The ODS score is the sum of all points, with a minimum of 0 point and a maximum possible of 31 points with higher scores meaning worse outcome.
Quality of life by the use of the Short Form (36) Health Survey (SF-36) questionnaire | At baseline and at 24-month
  Change from screening of each domain score and total score at 24-month. The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100 with lower scores = more disability, and higher scores = less disability
Description of device deficiency: inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance. Device deficiencies include malfunctions, use errors, and inadequate labelling. | During the surgical procedure
  Summarized and listed

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume MEURETTE, MD, Principal Investigator — CHU Nantes, France
Locations (3):
- France (3):
  - CHU Estaing, Clermont-Ferrand
  - CHU Nantes Hôtel Dieu, Nantes
  - Hôpital Haut-Lévèque- CHU de Bordeaux, Pessac

IPD SHARING:
Plan to Share IPD: No